CLINICAL TRIAL: NCT07027722
Title: Clinical Practices for Treating Severe Malaria Caused by P. Falciparum
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0066_SMIT
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Malaria, Falciparum; Plasmodium Falciparum; Antimalarials; Artemisinins; Treatment Outcome; Drug Therapy, Combination; Retrospective Studies; Hospitalization
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study looks at how doctors in three hospitals in France treat patients with a serious form of malaria caused by Plasmodium falciparum. It focuses on cases where the level of malaria parasites in the blood is 4% or higher. The study will compare how often a type of medicine called ACT (artemisinin-based combination therapy) is used on its own instead of the usual first-choice treatment (intravenous artesunate), and whether ACT works just as well. It will also check how well patients recover, whether they have complications, and how long they stay in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Diagnosis of Plasmodium falciparum malaria with a parasitemia level ≥ 4%.

Exclusion Criteria:

- Patients under 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (aged 18 years and older) who were hospitalized in one of the three participating centers over the past five years for Plasmodium falciparum malaria with a parasitemia level greater than or equal to 4%. These patients may or may not have presented with clinical signs of severity, and their treatment will have included either artemisinin-based combination therapy (ACT) or intravenous artesunate. Participants will be selected retrospectively from medical records based on these criteria.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients treated with artemisinin-based combination therapy (ACT) alone for Plasmodium falciparum malaria with parasitemia ≥4%. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France